CLINICAL TRIAL: NCT03617666
Title: AVENuE - Avelumab in the Frontline Treatment of Advanced Classical Hodgkin Lymphoma - a Window Study
Brief Title: Avelumab in the Frontline Treatment of Advanced Classical Hodgkin Lymphoma - a Window Study
Acronym: AVENuE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL /17/0192; 2018-002227-42 (EudraCT Number)
Record Dates: First submitted 2018-07-20; First posted 2018-08-06 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Hodgkin Lymphoma
Keywords: avelumab
MeSH Terms: conditions — Hodgkin Disease | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Avelumab (Experimental): Patients with newly diagnosed cHL will receive single agent avelumab in 2 cycles
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Patients with newly diagnosed cHL will receive 4 doses of single agent avelumab 10 mg/kg intravenously given every 2 weeks.
  Other Names: Bavencio

SUMMARY:
This is a phase II, non-randomised, multicentre study to assess the safety and efficacy of the PD-L1 inhibitor, avelumab, in a previously untreated fit population of high risk stage II, stage III and stage IV classical Hodgkin lymphoma.

DETAILED DESCRIPTION:
This phase II study investigates the safety and efficacy of the PD-L1 inhibitor, avelumab, in a previously untreated fit population of high risk stage II, stage III and stage IV classical Hodgkin lymphoma.

Patients with newly diagnosed high risk stage II, stage III or stage IV cHL staged by 18FDG-PET/CT will receive 4 doses of single agent avelumab every 2 weeks. After the 4th dose of avelumab patients will have a PET-CT scan. All patients will then receive 2 cycles of ABVD followed by a PET-CT scan and further treatment will be guided in a risk-adapted manner based on the results of the RATHL. That is, patients who achieve PET CMR (defined as Deauville score 1-3) will receive 4 cycles of AVD and will undergo a CT scan. Patients with Deauville score 4-5 will receive 4 cycles of BEACOPP-14 or 3 cycles of escalated BEACOPP (at Investigators discretion and as per standard local policy) and will then undergo a further PET scan. Patients who are Deauville score 1-3 at this point will receive 2 further cycles of BEACOPP-14 or 1 cycle of escalated BEACOPP (at Investigators discretion and as per standard local policy). Patients who are Deauville score 4-5 at this point will receive further treatment at Investigators discretion and as per standard local policy. Radiotherapy to sites of residual avidity, initial bulk or as part of salvage treatment, is recommended (but not mandated).

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated classical Hodgkin lymphoma
* High risk stage II (defined as stage IIB, presence of bulky disease, 3 or more sites of disease), stage III or IV as assessed by FDG-PET/CT
* ECOG performance status 0-1
* Adequate bone marrow function (Hb >80g/l, Platelets >75 x 10^9/l, neutrophils >1.0 x 10^9/l)
* Adequate liver function tests (ALT/AST <2.5 x ULN, total serum bilirubin level <1.5 x ULN)
* Creatinine clearance >50ml/min calculated by Cockroft-Gault formula
* Written informed consent
* Willing to comply with the contraceptive requirements of the trial
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Nodular lymphocyte predominant Hodgkin lymphoma
* Compressive symptoms due to disease (which may or may not be bulky). If there is evidence of compression of vital structures radiologically but the patient is asymptomatic, the case must be discussed with the TMG.
* Requirement for urgent treatment due to life-threatening complications of the disease
* Women who are pregnant or breastfeeding
* History of colitis, inflammatory bowel disease or pneumonitis
* Patients with autoimmune disorders excluding patients with vitiligo, diabetes mellitus type 1, hypo- and hyperthyroidism, coeliac disease not requiring immunosuppressive therapy
* Immunosuppressive therapy within the last 2 months, apart from inhaled, intranasal, topical corticosteroids or systemic corticosteroids at low doses (≤10mg prednisolone per day or equivalent - see steroid exception below)
* Prior history of solid organ or allogeneic haematopoietic stem cell transplant
* Positive serology for hepatitis B or C (unless due to vaccination), or hepatitis C RNA negative if hepatitis C antibody positive
* Known HIV infection
* Administration of a live vaccine within 30 days prior to study entry
* History of allergy to monoclonal antibodies, anaphylaxis or uncontrolled allergy
* Chemo- or radiotherapy within 15 days prior to registration. Corticosteroids permitted for disease control but must be weaned down to ≤10mg prednisolone per day or equivalent at least 7 days prior to starting avelumab - steroids may only be started for disease control after the baseline PET-CT
* Persisting toxicity (of >grade 1) related to prior therapy, however, alopecia, sensory neuropathy Grade <2, or other grade <2 not constituting a safety risk based on investigator's judgement are acceptable
* Major surgery within 4 weeks prior to registration
* Active infection requiring systemic therapy
* Myocardial infarction, unstable angina, coronary artery bypass graft, cerebrovascular accident or transient ischaemic attack within the past 6 months
* Non-haematological malignancy within the past 3 years (some exceptions apply)
* Previously treated haematological malignancy
* Any uncontrolled medical condition which can impair delivery of planned immunochemotherapy
* Patient not deemed suitable for ABVD/AVD/escalated-BEACOPP/BEACOPP-14

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 2 months (after first dose of avelumab)
  Overall response rate (complete metabolic response (CMR) and partial metabolic response (PMR)) after 2 months (4 doses) of single agent avelumab treatment

SECONDARY OUTCOMES:
Progression free survival | 1 year and 3 years (from date of registration)
  Progression free survival will be calculated from the date of registration until the date of progression.
Overall survival | 1 year and 3 years (from date of registration)
  Overall survival time will be calculated from the date of registration until the date of death.
Rates of adverse events with avelumab | 3 months (after first dose of avelumab)
  Safety and toxicity of avelumab, particularly autoimmune toxicity, as assessed by CTCAE v5.0
Rates of adverse events with ABVD/BEACOPP | 7 months (after commencing ABVD/BEACOPP)
  Safety and toxicity of subsequent ABVD/BEACOPP based chemotherapy, as assessed by CTCAE v5.0
Complete metabolic response rate | 2 months (after commencing ABVD)
  Complete metabolic response rate following 2 cycles of ABVD
Partial metabolic response rate | 2 months (after commencing ABVD)
  Partial metabolic response rate following 2 cycles of ABVD
Treatment compliance | 9 months (from the date of registration)
  Proportion of patients completing chemotherapy without delays/dose modifications and proportion of patients who have chemotherapy dose delay/modification.

OTHER OUTCOMES:
Correlate PET positive disease | End of trial (3 years)
  Correlate PET positive disease with histological evidence of disease on biopsy to establish biopsy negative PMR rate (subject to patient consent)
Correlate disease response | End of trial (3 years)
  Correlate disease response, as assessed by FDG-PET and histology, with serological markers, including serum TARC
Correlation between response to avelumab and biological parameter | End of trial (3 years)
  Evaluate the correlation between response to avelumab and biological parameters e.g. PD-1 expression on Reed Sternberg cells

CONTACTS AND LOCATIONS:
Overall Officials: Graham Collins, Principal Investigator — Churchill Hospital
Locations (11):
- Austin Health, Heidelberg, Victoria, Australia
- United Kingdom (10):
  - Heartlands Hospital, Birmingham
  - Beatson Hospital, Glasgow
  - Leicester Royal Infirmary, Leicester
  - St George's Hospital, London
  - Christie Hospital, Manchester
  - Norfolk and Norwich University Hospital, Norwich
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Royal Stoke University Hospital, Stoke
  - The Royal Marsden Hospital, Sutton, Sutton

IPD SHARING:
Plan to Share IPD: No